CLINICAL TRIAL: NCT00544544
Title: Riluzole in the Treatment of Bipolar Depression: A Study of the Association Between Clinical Response and Change in Brain Glutamate Levels as Measured by Proton Magnetic Resonance Spectroscopy
Brief Title: Riluzole in the Treatment of Bipolar Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Brian P. Brennan, MD, Associate Director of Translational Neuroscience Research, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-P-000751
Record Dates: First submitted 2007-10-12; First posted 2007-10-16 (Estimated); Results first posted 2010-08-18 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Bipolar Depression
Keywords: Bipolar; depression
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Riluzole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Riluzole (Experimental): Riluzole 50 mg twice daily for 2 weeks, increased to riluzole 50 mg in the morning and 100 mg in the evening for 1 week if tolerated, with a further increase to riluzole 100 mg twice daily if tolerated for 3 weeks.
  Interventions: Drug: Riluzole

INTERVENTIONS:
Drug: Riluzole — 50 mg twice daily for 2 weeks 50 mg in the morning and 100 mg in the evening for 1 week 100 mg twice daily for 3 weeks
  Other Names: Rilutek

SUMMARY:
Bipolar disorder is a common and often chronic and debilitating mental illness. The depressive phase of bipolar disorder contributes the largest portion of the disorder, and treatment resistant bipolar depression represents a significant public health problem. Recent research has suggested that bipolar depression is associated with elevated brain glutamate activity. We hypothesize that riluzole, a drug approved for ALS which inhibits glutamate activity, will lead to clinical improvement in patients with bipolar depression.

DETAILED DESCRIPTION:
We hypothesize that riluzole will lead to significant reduction in depressive symptoms as measured by the Hamilton Depression Rating Scale (HAM-D). Additionally, improvement in depressive symptoms will be associated with reduced glutamate levels in the anterior cingulate cortex, but not parieto-occipital cortex, both at day two and day 42.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18-65
* Meets DSM-IV criteria for Bipolar Disorder and is currently depressed
* Current score of >/= 18 on the Hamilton Depression Scale

Exclusion Criteria:

* Active psychotic/manic symptoms
* Lifetime history of schizophrenia or obsessive compulsive disorder
* Clinically significant medical disease
* Women who are pregnant or lactating and women who are not using a medically accepted method of contraception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-06; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dost Ongur, M.D, Ph.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

REFERENCES:
- [Result] Brennan BP, Hudson JI, Jensen JE, McCarthy J, Roberts JL, Prescot AP, Cohen BM, Pope HG Jr, Renshaw PF, Ongur D. Rapid enhancement of glutamatergic neurotransmission in bipolar depression following treatment with riluzole. Neuropsychopharmacology. 2010 Feb;35(3):834-46. doi: 10.1038/npp.2009.191. Epub 2009 Dec 2. PMID 19956089

RESULTS

PARTICIPANT FLOW:
Groups:
- Riluzole: Riluzole 100-200 mg/day
Period: Overall Study
Arm/Group | Riluzole
Started | 14
Completed | 11
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Riluzole
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Depression Rating Scale
Description: The Hamilton Depression rating Scale is a clinician-rated scale that measures the severity of depression symptoms using 21 items. Minimum score is zero and maximum score is 65. Higher scores indicate more severe depressive symptoms.
Time Frame: Baseline (week 0) - week 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Riluzole
Number analyzed (Participants) | 14
units on a scale | -12.6 [-16.5 to -8.6]
Statistical Analysis 1: Comparison: Riluzole; Test type: Superiority or Other; p < .001, Mixed Models Analysis

2. Secondary Outcome: Montgomery Asberg Depression Rating Scale
Description: The Montgomery-Asberg Depression Rating Scale is a clinician-rated scale that measures the severity of depression symptoms. The 10 items measured are apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Minimum score is zero and maximum score is 60. Higher scores represent more severe depressive symptoms.
Time Frame: Baseline (week 0) - week 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Riluzole
Number analyzed (Participants) | 14
units on a scale | -13.0 [-18.0 to -8.0]
Statistical Analysis 1: Comparison: Riluzole; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

3. Secondary Outcome: Young Mania Rating Scale
Description: The Young Mania Rating Scale is a clinician-rated scale that measures the severity of mania symptoms. The 11 items measures are elevated mood, increased motor activity, sexual interest, sleep, irritability, speech, language-thought disorder, thought content, aggressive behavior, appearance, and insight. Minimum score is zero and maximum score is 60. Higher scores represent more severe mania symptoms.
Time Frame: Baseline (week 0) - week 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Riluzole
Number analyzed (Participants) | 14
units on a scale | -0.6 [-2.0 to 0.7]
Statistical Analysis 1: Comparison: Riluzole; Test type: Superiority or Other; p = 0.38, Mixed Models Analysis

4. Secondary Outcome: Clinical Global Impression Scale
Description: The Clinical Global Impression Scale is a clinician-rated scale that evaluates the severity of illness at the time of assessment. The score ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Baseline (week 0) - week 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Riluzole
Number analyzed (Participants) | 14
units on a scale | -1.6 [-2.4 to -0.8]
Statistical Analysis 1: Comparison: Riluzole; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Riluzole
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 14/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riluzole (N=14)
nausea (Gastrointestinal disorders) | 6 (6)
headache (Nervous system disorders) | 4 (4)
diarrhea (Gastrointestinal disorders) | 4 (4)
insomnia (Nervous system disorders) | 4 (4)
constipation (Gastrointestinal disorders) | 3 (3)
sedation (Nervous system disorders) | 3 (3)
neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
dizziness (Nervous system disorders) | 2 (2)
dry mouth (General disorders) | 2 (2)
back pain (Musculoskeletal and connective tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No